CLINICAL TRIAL: NCT04961086
Title: Effect of Consumption of Energy Drinks on Hemodynamics, Blood Glucose, Short Term Memory, Vigilance and Perception in Healthy Adults
Brief Title: Health Effect of Energy Drink Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, SM Ashraf Jahangeer, Doctor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHS001
Record Dates: First submitted 2021-06-28; First posted 2021-07-14 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Blood Pressure; Blood Glucose, High; Cognitive Change
Keywords: energy drink; hemodynamics; memory; stroop test
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- energy drink arm (Experimental): an open label branded energy drink which contains any one or more of the following ingredients: caffeine, ginseng, taurine
  Interventions: Other: energy drink
- tea 5gm sugar arm (Active Comparator): the usual easily available black tea with sugar 5 grams, and milk
  Interventions: Other: energy drink

INTERVENTIONS:
Other: energy drink — An easily available 250 ml branded energy drink will be randomized to the partcipants after informed consent. Before and thirty minutes after drinking the given energy drink the participant cognition, heart rate, blood pressure and blood glucose will be measured.

SUMMARY:
Energy drinks consumption has varied effects on the hemodynamic, blood glucose levels, brain functions and memory. The use of energy drinks is pervasive and especially young adults consume it often as binge drinking. The negative health effects of excessive use of energy drinks has been reported in the scientific literature. Often energy drinks are consumed to enhance alertness and cognition improvement. In this trial, the investigators intend to compare the effects of a widely available energy drink brand in the country with the usual black tea with 5gm sugar and milk. The aims of this study is:

1. To determine the effect of consumption of energy drinks on hemodynamics parameters.
2. To determine the effect of consumption of energy drinks on short term memory
3. To determine the effect of consumption of energy drinks on vigilance in adults
4. To determine the effect of consumption of energy drinks on blood glucose in adults
5. To analyze the effect of energy drink on perception in adults

DETAILED DESCRIPTION:
The participants will be halved in two groups: control group (consuming tea with 5gm of sugar only) and experimental group (consuming energy drinks only) to acquire data regarding fluctuations in hemodynamic parameters including heart rate (HR) and blood pressure (BP)-systolic and diastolic (SBP and DBP) by measuring them before and after 30 minutes of the consumption of tea with 5gm of sugar or energy drink in control or experimental groups. In addition blood glucose level will be monitored in both the groups via glucometer before and after. Reactions of energy drinks in comparison to tea on their respective groups will also be analyzed by help of a stroop test (where the name of the color itself does not match the ink of the color in which it is printed) for understanding its impact on cognitive strengths and on memory by a minor sequence learning game controlled by time lapse. After these interventions participants will be requested to fill out the questionnaire.

The investigatorsare aiming for a sample size of 76 participants, 38 in each of the two groups.

Data will be entered and analyzed in Statistical Package for the Social Sciences version 20 or above. Mean and SD will be calculated for variables such as age, weight, blood pressure (Systolic and Diastolic) and heart rate, blood glucose and Stroop Test score. For qualitative variables such as sex, co morbidity e.g. heart disease, hypertension, family history will be presented as absolute frequencies and proportions. The hemodynamic parameters will be recorded before and after consumption of energy drinks in the intervention and the control group. Independent samples student t-test will be used to compare mean values of hemodynamic parameter between intervention and control group. Significance level of 5% will be set for the study keeping power at 80%.

ELIGIBILITY:
Inclusion Criteria

* Adult volunteers aged between 18-30 years
* Either gender
* Willing to participate

Exclusion Criteria:

* Known cardiovascular diseases
* Under any medication
* Known Diabetes mellitus or any other chronic disease
* Pregnancy or lactation
* History of neurological disorders
* History of regular alcohol consumption

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | half hour post consumption
  before and after consumption of the energy drink or the tea both systolic and diastolic blood pressures will be measured as per international guidelines for measuring BP
Change in heart rate | half hour post consumption
  before and after consumption of the energy drink or the tea heart rate will be measured as per international guidelines
Change in blood glucose | half hour post consumption
  before and after consumption of the energy drink or the tea blood glucose levels will be measured as per international guidelines
Change in short-term memory and vigilance | half hour post consumption
  before and after consumption of the energy drink or the tea short term memory functions will be measured using color sequence game. We will use STROOP test to assess vigilance

SECONDARY OUTCOMES:
perceptions and knowledge of participants about energy drinks | within one hour of consumption of the energy drink or the active comparator
  simple questions from the participants about the effects and composition of energy drinks

CONTACTS AND LOCATIONS:
Overall Officials: Syed Muhammad Ashraf Jahangeer, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, None Selected, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nowak D, Jasionowski A. Analysis of the Consumption of Caffeinated Energy Drinks among Polish Adolescents. Int J Environ Res Public Health. 2015 Jul 10;12(7):7910-21. doi: 10.3390/ijerph120707910. PMID 26184263
- [Result] Nowak D, Goslinski M, Nowatkowska K. The Effect of Acute Consumption of Energy Drinks on Blood Pressure, Heart Rate and Blood Glucose in the Group of Young Adults. Int J Environ Res Public Health. 2018 Mar 19;15(3):544. doi: 10.3390/ijerph15030544. PMID 29562659
- [Result] Wesnes KA, Brooker H, Watson AW, Bal W, Okello E. Effects of the Red Bull energy drink on cognitive function and mood in healthy young volunteers. J Psychopharmacol. 2017 Feb;31(2):211-221. doi: 10.1177/0269881116681459. Epub 2016 Dec 14. PMID 28168925
- [Result] Buckenmeyer PJ, Bauer JA, Hokanson JF, Hendrick JL. Cognitive influence of a 5-h ENERGY(R) shot: Are effects perceived or real? Physiol Behav. 2015 Dec 1;152(Pt A):323-7. doi: 10.1016/j.physbeh.2015.09.003. Epub 2015 Sep 21. PMID 26394126
- [Result] Smith AP, Richards G. Energy drinks, caffeine, junk food, breakfast, depression and academic attainment of secondary school students. J Psychopharmacol. 2018 Aug;32(8):893-899. doi: 10.1177/0269881118783314. Epub 2018 Jun 27. PMID 29947575
- [Result] Brothers RM, Christmas KM, Patik JC, Bhella PS. Heart rate, blood pressure and repolarization effects of an energy drink as compared to coffee. Clin Physiol Funct Imaging. 2017 Nov;37(6):675-681. doi: 10.1111/cpf.12357. Epub 2016 Mar 1. PMID 26931509